CLINICAL TRIAL: NCT05682482
Title: A National Randomized Placebo-controlled Double-blind Multicenter Trial of LT4/LT3 Combination Therapy in Patients with Autoimmune Hypothyroidism: the T3-4-Hypo Trial.
Brief Title: LT4/LT3 Combination Therapy Versus LT4 Monotherapy in Patients with Autoimmune Hypothyroidism.
Acronym: T3-4-Hypo
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M. Medici (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); ACE Pharmaceuticals BV (Other)
Responsible Party: Sponsor-Investigator, M. Medici, Dr. M. Medici, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL74281.078.21
Record Dates: First submitted 2021-11-01; First posted 2023-01-12 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-08

CONDITIONS: Autoimmune Hypothyroidism
Keywords: Triiodothyronine; Quality of life; Persistent complaints
MeSH Terms: conditions — Hypothyroidism, Autoimmune | interventions — Triiodothyronine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LT4/LT3 combination therapy (Active Comparator): The intervention group is treated with once daily a LT4 tablet and twice daily a LT3 tablet with a LT4:LT3 ratio 16:1.
  Interventions: Drug: LT3 (liothyronine)
- LT4/placebo therapy (Placebo Comparator): The control group is treated with once daily a LT4 tablet and twice daily a placebo tablet.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LT3 (liothyronine) — Addition of liothyronine (LT4/LT3 combination therapy) in patients with persistent tiredness on LT4 monotherapy. To investigate whether addition of LT3 is effective in relieving tiredness.
  Other Names: Intervention group LT4/LT3 combination therapy
  Arms: LT4/LT3 combination therapy
Drug: Placebo — Addition of placebo (LT4 monotherapy) in patients with persistent tiredness on LT4 monotherapy.
  Other Names: Control group LT4/placebo therapy
  Arms: LT4/placebo therapy

SUMMARY:
Hypothyroidism is common, affecting 5% of the general population, for which levothyroxine (LT4) monotherapy is the standard treatment. Despite normalized serum thyroid hormone levels, 10-15% of LT4 treated patients have various persistent complaints, the most important of which is tiredness. This could be explained by the fact that physiological T4/T3 ratios cannot be reached with LT4 monotherapy, as in a healthy individual T3 is not only derived from T4/T3 conversion but is also directly produced by the thyroid itself. Studies have reported contradicting results as to whether addition of liothyronine (LT4/LT3 combination therapy) in patients with persistent tiredness on LT4 monotherapy is effective or not. Studies have suggested higher effectiveness in patients carrying genetic variation in the type 2 deiodinase (DIO2-rs225014) and monocarboxylate transporter 10 (MCT10-rs17606253) genes.

Objective: To investigate whether addition of liothyronine (LT4/LT3 combination therapy) in in patients with persistent tiredness on LT4 monotherapy is effective or not in relieving tiredness.

DETAILED DESCRIPTION:
After obtaining informed consent we will enroll patients with autoimmune hypothyroidism and persistent tiredness despite normalized TSH levels on LT4 monotherapy. A general physical examination will be performed, and in- and exclusion criteria will be checked. This also includes an ECG to prevent including patients with a functional or structural abnormal heart. The study will start with a run-in period, during which all patients switch to blinded generic LT4, which is produced and distributed by the trial pharmacy. This is because there are seven LT4 preparations available in the Netherlands with different pharmacokinetic properties, which would otherwise introduce substantial bias. Previous research has shown that 36% of patients need dose adjustments when switching to other LT4 preparations. Therefore, serum TSH levels are measured every 8 weeks, and medication dosages adjusted if needed, in order to obtain normal serum TSH levels, defined as TSH levels within the assay-specific reference range. For trial feasibility, patients will be excluded from this study and referred back to their referring physician when a normal TSH cannot be reached with a maximum of two dose adjustments. Once a normal TSH has been measured, the final run-in TSH measurement will be performed 8 weeks later. This is because we want to ensure that we only enroll patients with a stable (i.e. normal) TSH on a stable dose of generic LT4, as recent dose adjustments could otherwise impact the tiredness questionnaire scores at the start of the RCT. This TSH measurement will be combined with a repeat ECG and the patient will be asked whether tiredness with a large negative impact on daily life is still present. Patients will enter Stage 2 (RCT) when they have a normal TSH, no ECG abnormalities, and indicate they have persistent tiredness. Patients not fulfilling these criteria will be excluded from this study and referred back to their referring physician. The expected duration of the run-in period will be 4-8 months, depending on the number of dose adjustments.

Stage 2 includes a 1-year double-blind randomized placebo-controlled trial comparing LT4/LT3 with LT4/placebo treatment. At baseline, patients are randomized to either LT4/LT3 or LT4/placebo treatment. Serum TSH levels are measured at every visit, and medication dosages adjusted if needed, with the goal to normalize serum TSH levels, defined as TSH levels within the assay-specific reference range. Patients are excluded and referred back to their referring physician in case a normal TSH cannot be reached with the available study medication dosages (62,5 - 237,5 µg LT4 monotherapy dose). Visits will take place at baseline, and weeks 8, 16, 26, 39 and 52. The density of visits is higher at the beginning as this is the period when dose adjustments are particularly expected. At every visit, patients are asked to complete questionnaires on thyroid related complaints and quality of life (ThyPRO), general quality of life (EuroQoL-5D-5L and EuroQoL-5D-VAS), medical consumption (iMCQ) and productivity losses (iPCQ). At baseline and 52 weeks, additional blood will also be drawn to determine genetic variants, (thyroid hormone) metabolites and collect material for biobanking, as these data will be key to identify subgroups who are likely to respond to LT4/LT3 combination therapy. Although we do not expect any detrimental effects of these low physiological LT3 dosages, and previous studies neither reported any detrimental effects, we will explore the effects of LT4/LT3 combination therapy on the most important thyroid hormone target organs (bone, cardiovascular, metabolic and brain). This will improve communication between medical professionals and patients, providing them with comprehensive information on the balance between the potential benefits and harms of combination therapy vs monotherapy and will enable shared-decision making that better addresses individual needs of patients. For bone, serum bone markers will be determined at baseline and 52 weeks, and DXA scans will be performed at baseline and 52 weeks in a subgroup of 200 individuals. For cardiovascular and metabolic endpoints, blood pressure, pulse rate, weight, and waist circumference are measured at every visit. Fat percentages will be assessed on the beforementioned DXA scans. A repeat ECG will be performed at 52 weeks. To objectively explore effects on neurocognitive function, next to the subjective ThyPRO questionnaire scores, neurocognitive tests will be performed in a subgroup of 200 patients at baseline and 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with overt or subclinical primary hypothyroidism 18 years or older.*
* LT4 monotherapy for at least 6 months.
* LT4 monotherapy dose of 75-225 microg, with at least a dose of 1.2 microg/kg.
* TSH levels within the assay-specific reference ranges for at least 3 months.
* Severe tiredness with a large negative impact on daily life for at least 6 months, with or without other persisting complaints. This is based on the patient's own experience, without judgment of the treating physician.
* Sufficiently fluent in Dutch and able to read Dutch.

  * Thyroid peroxidase (TPO) and/or thyroglobulin (Tg) antibody positivity is not a requirement as these have frequently not been determined. Instead, we ensure that we only include patients with autoimmune hypothyroidism by excluding other causes of hypothyroidism (see exclusion criteria).

Exclusion Criteria:

* Congenital hypothyroidism, hypothyroidism after (sub)acute thyroiditis*, secondary (central) hypothyroidism
* Thyroid surgery, radioactive iodine treatment, or head and/or neck radiotherapy.
* Use of thyroid interfering drugs (current/past use of amiodarone, immunotherapy, tyrosin kinase inhibitors, interferon, or lithium and current use of oral or iv corticosteroids or dopamine).
* Current psychiatric disease treated at a "gespecialiseerde GGZ instelling"**
* Clinical diagnosis of dementia.
* Pregnancy, breastfeeding or wish to become pregnant within 2 years.
* Women of reproductive age not using adequate contraception, who are not sterilized and do not have a sterilized partner. Adequate contraceptives include the contraceptive pill, patch, injection, implant, intrauterine device or system, vaginal ring, diaphragm or cap, and condom.
* Clinically relevant functional or structural abnormal heart (e.g., cardiomyopathy or valve disease)
* Recent acute coronary syndrome or unstable angina pectoris (<4 weeks)
* Current/past atrial fibrillation
* Current conduction disorder on ECG (i.e, QRS>120 ms or prolonged QTc (women≥460 ms and men≥450 ms)).
* Frequent ventricular extrasystole (=doublet, trigeminy, bigeminy or (non-sustained) ventricular tachycardia) in the past or on current ECG.
* Other obvious medical explanation for tiredness (e.g. end-stage renal disease, anemia, COPD stage IV, cancer, etc.)
* Other obvious major life event explanation for tiredness (e.g., mourning, loss of job)

  * Postpartum thyroiditis is not an exclusion criterium.
  * Treatments of mild non-complex psychological/psychiatric complaints are done in the " basis GGZ", e.g. consisting of conversations with a psychologist or psychotherapist, or via internet (e-health). "Gespecialiseerde GGZ" encompasses treatments of more severe psychological/psychiatric complaints. (link: Basis GGZ en gespecialiseerde GGZ | Geestelijke gezondheidszorg (GGZ) | Rijksoverheid.nl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline to 52 weeks in the ThyPRO tiredness subscale scores. | 52 weeks
  Thyroid specific Patient Reported Outcome (ThyPRO) questionnaire, with the tiredness subscale ranging from 0-100 (higher scores indicate a worse outcome).
  ThyPRO Questionnaires will be performed at every RCT visit.
Effect sizes in genetic subgroups | 52 weeks
  In case it is confirmed that LT4/LT3 combination therapy reduces tiredness compared to LT4 treatment alone, we will simultaneously investigate whether effect sizes are higher in patients with genetic variation in the type 2 deiodinase (DIO2-rs225014) and effect sizes are higher in patients with genetic variation in the monocarboxylate transporter 10 (MCT10-rs17606253), ensuring control of the study-wise type 1 error (of 5% two-sided) across these three main questions.

SECONDARY OUTCOMES:
Mean change from baseline to 52 weeks in the ThyPRO-39 composite scale* scores. | 52 weeks
  The Composite scale is based on 22 items from the Tiredness, Cognition, Anxiety, Depressivity, Emotional Susceptibility, Impaired Social life, Impaired Daily Life and Overall QoL subscales of the Thyroid specific Patient Reported Outcome (ThyPRO) questionnaire, with each subscale ranging from 0-100 (higher scores indicate a worse outcome).
  The ThyPRO questionnaire will be performed at every RCT visit.
Change from baseline to 52 weeks in the ThyPRO tiredness subscale scores ≥ minimal important difference (=14.3). | 52 weeks
  Thyroid specific Patient Reported Outcome (ThyPRO) questionnaire, with the tiredness subscale ranging from 0-100 (higher scores indicate a worse outcome).
  ThyPRO Questionnaires will be performed at every RCT visit.
Mean change from baseline to 52 weeks in the ThyPRO tiredness subscale scores in participants with a baseline score > 57 (= population mean, unpublished results; personal communication with Dr T Watt, developer of the ThyPRO questionnaire). | 52 weeks
  Thyroid specific Patient Reported Outcome (ThyPRO) questionnaire, with the tiredness subscale ranging from 0-100 (higher scores indicate a worse outcome).
  ThyPRO Questionnaires will be performed at every RCT visit.
Mean change from baseline to 52 weeks in the ThyPRO tiredness subscale scores in participants with a normal-range TSH level at 52 weeks. | 52 weeks
  Thyroid specific Patient Reported Outcome (ThyPRO) questionnaire, with the tiredness subscale ranging from 0-100 (higher scores indicate a worse outcome).
  ThyPRO Questionnaires will be performed at every RCT visit.
Determinants of the effects of LT4/LT3 combination therapy on tiredness. | 52 weeks
  Thyroid specific Patient Reported Outcome (ThyPRO) questionnaire, with the tiredness subscale ranging from 0-100 (higher scores indicate a worse outcome).
  ThyPRO Questionnaires will be performed at every RCT visit.
The (determinants of the) effects of LT4/LT3 combination therapy compared to LT4 therapy alone on other thyroid related complaints and quality of life. | 52 weeks
  Thyroid specific Patient Reported Outcome (ThyPRO) questionnaire, with the subscales ranging from 0-100 (higher scores indicate a worse outcome).
  ThyPRO Questionnaires will be performed at every RCT visit.
Number of adverse events in the LT4/LT3 combination therapy compared to the LT4 monotherapy groups. | 52 weeks
  AEs are defined as any undesirable experience occurring to a subject during the study, whether or not considered related to the investigational product / trial procedure. All following AEs according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be recorded, for which we also refer to the SmPCs for LT4 and LT3:
  * Hyperthyroidism (endocrine disorders subgroup)
  * Hypothyroidism (endocrine disorders subgroup)
  * All cardiac disorders subgroups
  * Erythroderma, rash and urticaria (skin and subcutaneous disorders subgroups)
  All other AEs will be recorded from CTCAE v 5.0 grade 3 onwards (= severe or medically significant but not immediately life-threatening).

CONTACTS AND LOCATIONS:
Overall Officials: Marco Medici, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (19):
- Netherlands (19):
  - Flevoziekenhuis, Almere Stad
  - Amsterdam UMC - Location AMC, Amsterdam
  - Gelre ziekenhuizen, Apeldoorn
  - Rijnstate, Arnhem
  - Amphia ziekenhuis, Breda
  - Van Weel-Bethesda Hospital, Dirksland
  - Albert Schweitzer Hospital, Dordrecht
  - Treant, Emmen
  - Admiraal de Ruyter Hospital, Goes
  - University Medical Center Groningen, Groningen
  - Saxenburgh MC, Hardenberg
  - Radboudumc, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - Maasstad Hospital, Rotterdam
  - Franciscus Gasthuis & Vlietland, Schiedam
  - Zuyderland, Sittard
  - University Medical Center Utrecht, Utrecht
  - Maxima Medical Center, Veldhoven
  - Vie Curie MC, Venlo

IPD SHARING:
Plan to Share IPD: Yes
A subset of the final data will be made available after an embargo period upon request. Most likely aggregated and filtered in order to maintain anonimity of individual patient data.
  The choice of online repository still has to be made.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: six months after database lock
Access Criteria: Upon request to the Principal investigator, with a sufficiently substantiated study proposal.

REFERENCES:
- [Derived] Phan GQ, Yavuz S, Stamatouli AM, Madan R, Chen S, Grover AC, Nilubol N, Bedoya P, Trankle C, Markley R, Abbate A, Celi FS. A feasibility double-blind trial of levothyroxine vs. levothyroxine-liothyronine in postsurgical hypothyroidism. Front Endocrinol (Lausanne). 2025 Mar 10;16:1522753. doi: 10.3389/fendo.2025.1522753. eCollection 2025. PMID 40130156
- See also: Trial website — http://www.t3-4-hypotrial.nl